CLINICAL TRIAL: NCT00297713
Title: A Phase II, Multi-Center, Multi-Dose, Randomized, Open-Label, Parallel Group Study of an Extended-Release, Crystalline Formulation of Recombinant Human Growth Hormone (ALTU-238) in Growth Hormone Deficient Adults to Determine Pharmacokinetics, Pharmacodynamics, and Drug Safety
Brief Title: Study of an Extended-Release, Crystalline Formulation of Recombinant Human Growth Hormone (ALTU-238) in Growth Hormone Deficient Adults to Determine Pharmacokinetics, Pharmacodynamics, and Drug Safety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altus Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230-00009
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2006-12-13 (Estimated); Status verified 2006-12

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

INTERVENTIONS:
Drug: ALTU-238

SUMMARY:
ALTU-238 is a long acting crystalline formulation of recombinant human growth hormone (rhGH) that is being developed for the treatment of growth hormone deficiency in adults and children. ALTU-238 is designed to require fewer injections than the currently available formulations of rhGH.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone deficient men and women ages 18-60 years with a hypothalamic and/or pituitary structural lesion or longstanding idiopathic GHD
* Growth hormone deficiency as determined by pituitary testing within the last five years by either of the two following tests:

  1. Insulin hypoglycemia (glucose < 50 mg/dL) with maximum GH < 5 ng/mL (5 µg/L) by radioimmunoassay or < 2.5 µg/L, if measured by immunoradiometric assay
  2. Arginine-GHRH infusions with maximum GH < 5 ng/mL (5 µg/L) or < 2.5 µg/L, if measured by immunoradiometric assay
* Women must be of non-child bearing potential (hysterectomy, tubal ligation, or IUD are acceptable) during the three months prior to entering the study, or post-menopausal (no menses for one year or more), or six to twelve months without menses and β-estradiol levels < 20 pg/mL
* Glucocorticoid use is allowed provided the subject has been on physiologic (<7.5 mg prednisone or equivalent/day) replacement doses for at least 3 months
* Free thyroxine (T4) within the normal range at Screening. If the subject is receiving thyroid hormone replacement therapy, the dose must be stable for at least 6 weeks prior to Screening
* Willing and able to provide written informed consent
* BMI 20 - 36 kg/m2

Exclusion Criteria:

* Any previous or ongoing clinically significant illness that, in the opinion of the investigator, could prevent the subject from completing the study
* Any history of cancer within the past 5 years, except for dermal squamous and basal cell carcinoma with documented 6-month remission. Subjects with a more recent history of successfully treated cervical carcinoma in situ will not be excluded provided there is documented 12-month remission
* BMI <20 or >36 kg/m2
* Any allergic or abnormal reaction to human growth hormone
* Inability of the subject to discontinue use of their regularly prescribed human growth hormone treatment from six weeks prior to Day -1 through the completion of the study
* Serum creatinine > 1.4 mg/dL
* Hypocalcemia or hypercalcemia from any cause
* Hyperparathyroidism, osteomalacia or any other disorder which may affect bone and bone markers including the use of bisphosphonates or other medications for osteoporosis
* Participation in another clinical trial 30 days prior to screening
* Demonstrated inability to comply with protocol requirements (e.g. uncooperative attitude, inability to return for follow-up visits, history of medical non-compliance, and/or poor likelihood of completing the study)
* Blood donation within 56 days of the screening visit
* Plasma donation within seven days of the screening visit
* Positive serum pregnancy test
* Women of child bearing potential
* Abuse of alcohol; to be determined by principal investigator
* Abuse of prescription or illicit drugs; to be determined by principal investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - University of Texas Medical Branch, Galveston, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas